CLINICAL TRIAL: NCT06071767
Title: A Phase I/IIa Randomized, Placebo-Controlled Trial of Conserved-Mosaic T-cell Vaccine in a Regimen With Vesatolimod and Broadly Neutralizing Antibodies in Adults Initiated on Suppressive Antiretroviral Therapy During Acute HIV-1
Brief Title: Evaluation of Safety, Immunogenicity and Efficacy of a Triple Immune Regimen in Adults Initiated on ART During Acute HIV-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Oxford (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5374; 12025 (Other: DAIDS-ES ID); HIV-CORE 009 (Other: University of Oxford clinical program for developing T-cell vaccines for conserved HIV protein regions)
Record Dates: First submitted 2023-09-05; First posted 2023-10-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection
Keywords: Suppressive Antiretroviral Therapy; HIV; Acute HIV-1; HIV vaccine; T-cell vaccine; Therapeutic T-cell vaccine; ChAdOx1; MVA; Conserved region vaccine; HIVconsvX; Toll-like receptor 7 agonist; TLR7; Broadly neutralizing antibody; Antibodies; HIV antibody; HIV Broadly neutralizing antibody
MeSH Terms: interventions — vesatolimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs (Experimental)
  Interventions: Biological: ChAdOx1.tHIVconsv1; Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv3; Biological: MVA.tHIVconsv4; Drug: Vesatolimod (VES); Drug: GS-5423; Drug: GS-2872
- Arm B: Placebos for vaccines, vesatolimod and bnAbs (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ChAdOx1.tHIVconsv1 — Administered as 0.4 mL intramuscularly (IM) at Week 0
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Biological: ChAdOx1.HIVconsv62 — Administered as 0.3 mL IM at Week 0
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Biological: MVA.tHIVconsv3 — Administered as 0.3 mL IM at Week 4
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Biological: MVA.tHIVconsv4 — Administered as 0.5 mL IM at week 4
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Drug: Vesatolimod (VES) — VES 6 mg administered orally once every 2 weeks for two doses, then VES 8 mg once every 2 weeks for 8 doses. Dose escalation may be held or the 8 mg dose may be reduced for intolerability for weeks 6 through 24.
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Drug: GS-5423 — Administered via intravenous (IV) infusion at week 7
  Other Names: 3BNC117-LS; Teropavimab
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Drug: GS-2872 — Administered via IV infusion at week 7
  Other Names: 10-1074-LS; Zinlirvimab
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Biological: MVA.tHIVconsv4 — Administered 0.5 mL IM at week 60
  Arms: Arm A: Active ChAdOx1 and MVA/HIVconsvX vaccines, vesatolimod and bnAbs
Biological: Placebo — Placebos for vaccines, VES, and bnAbs
  Arms: Arm B: Placebos for vaccines, vesatolimod and bnAbs

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of therapeutic vaccination with chimpanzee adenovirus ChAdOx1- and poxvirus modified vaccinia Ankara (MVA)-vectored conserved mosaic T-cell vaccines in a sequential regimen with the toll-like receptor 7 (TLR7) agonist vesatolimod (VES) and two broadly neutralizing antibodies (bNAbs) compared to placebo, to induce HIV-1 control during analytic treatment interruption (ATI).

DETAILED DESCRIPTION:
A5374 is a phase I/IIa randomized, two-arm, double-blind placebo-controlled, multi-step strategy trial to evaluate safety and efficacy of therapeutic vaccination with chimpanzee adenovirus ChAdOx1- and poxvirus modified vaccinia Ankara (MVA)-vectored conserved mosaic T-cell vaccines in a sequential regimen with the toll-like receptor 7 (TLR7) agonist vesatolimod (VES) and two broadly neutralizing antibodies (bNAbs) of the CD4 binding site and V3-loop base classes in individuals with HIV-1 who started suppressive antiretroviral therapy (ART) during acute HIV-1.

Participants will be screened for eligibility and have a pre-entry visit. After determination of eligibility, participants will be randomized prior to entry to either the active intervention arm (Arm A) or the placebo arm (Arm B) in a 2:1 ratio.

The study consists of four steps including an analytical treatment interruption (ATI).

* Step 1: Study Intervention and ART (67 weeks)
* Step 2: Analytic Treatment Interruption (up to 24 weeks)
* Step 3: ART Restart (24 weeks)
* Step 4: Continuation of ATI (up to 24 weeks)

Each participant will complete Step 1 and Step 2. At the end of Step 2, participants who have experienced virologic rebound will enter Step 3 and resume ART. Participants who did not meet ART restart criteria after 24 weeks in Step 2 will enter Step 4 for an extended ATI.

Each participant will be enrolled for up to approximately 110 weeks. The total time on study for each participant is dependent on the time spent in the treatment interruption steps (Step 2 and 4).

ELIGIBILITY:
Inclusion Criteria

* Provision of written informed consent.
* History of Initiation of combination ART within 90 days of acute HIV diagnosis
* On ART for at least 12 months with no known ART interruption >28 consecutive days within 12 months prior to Step 1 Study Entry
* ART with an integrase inhibitor-based regimen with two NRTIs or dolutegravir/lamivudine regimen for at least 6 weeks prior to Study Entry.
* Willingness to participate in the ATI and willingness to restart ART according to study guidelines.
* Willingness to adhere to protocol therapy and complete all study visits.
* Weight ≥50 kg and ≤150 kg at Screening.
* CD4 cell count ≥500 cells/mm3 obtained within 60 days prior to Study Entry.
* HIV-1 RNA <50 copies/mL (or below the assay limit of quantification if local assay lower limit of quantification is >50 copies/mL) for at least 1 year and within 60 days prior to Study Entry.
* Select laboratory results within 60 days of study entry
* For cisgender women and transgender men of reproductive potential, negative urine or serum pregnancy test within 48 hours prior to or at study Entry.
* Participants who are able to become pregnant and who are engaging in sexual activity that could lead to pregnancy must agree to use two methods of contraception, one of which must be a highly effective methods for contraception. Barrier methods of contraception are required for the second method of contraception.
* Availability of results of HLA typing (required for randomization).
* Completion of pre-entry leukapheresis or LVBD.

Exclusion Criteria

* Currently pregnant or breastfeeding or planning to become pregnant during study participation.
* Prior receipt of anti-HIV broadly neutralizing antibody therapy.
* Receipt of any non-HIV monoclonal antibody therapy within 1 year prior to study entry.
* Prior receipt of a latency-reversing agent (LRA).
* Receipt of HIV-1 or other investigational vaccines within 6 months prior to Study Entry.
* Receipt of a live-virus vaccine within 60 days or any vaccination within 14 days prior to Study Entry.
* Receipt of any simian adenovirus-vectored vaccine (e.g., anti-COVID-19 AZD1222) within 12 months prior to Step 1 Study Entry.
* Known allergy/sensitivity or any hypersensitivity to components of study treatments or their formulations.
* Known severe chicken egg allergy.
* Known history of a severe reaction or anaphylaxis to prior vaccinations or antibody preparations (e.g., intravenous immunoglobulin).
* Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity).
* Any history of anaphylaxis and related symptoms such as hives, respiratory difficulty, or angioedema.
* Previous or current history of bleeding factor deficiency, coagulopathy or platelet disorder or on chronic anticoagulation.
* History of inflammatory neurologic diseases.
* History of pregnancy, head trauma or major surgery within 90 days prior to Step 1 Study Entry.
* History of use of any immunomodulatory medications within the 6 months prior to Step 1 Study Entry.
* Significant serious skin disease, such as but not limited to active rash, eczema, psoriasis, or urticaria.
* Autoimmune disease (e.g., lupus, multiple sclerosis, and others) requiring ongoing immunosuppression.
* Known history of CDC Stage 3 opportunistic infection (OI).
* Any history of an HIV-associated malignancy.
* Known or suspected active or untreated latent Mycobacterium tuberculosis infection.
* Active or recent non-HIV-associated malignancy.
* Serious illness requiring systemic treatment and/or hospitalization within 90 days prior to study entry.
* Known resistance to one or more drugs in two or more ARV drug classes.
* History of or current clinical atherosclerotic cardiovascular disease
* Current advanced liver disease.
* Use of complementary or alternative medicines within 14 days prior study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-04-29 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any serious adverse event (AE), Grade 3 or higher AE, or AE that leads to permanent discontinuation of study treatment regardless of grade, that is related to ChAdOx1-MVA/HIVconsvX vaccines, vesatolimod, GS-5423 or GS-2872 | Week 0 to Week 64
Proportion of participants with viral control during an ATI defined as remaining off ART with HIV-1 RNA <1,000 copies/mL at Week 16 following ATI. | Week 0 to Week 16 on Step 2

SECONDARY OUTCOMES:
Change in cell-associated HIV-1 RNA and DNA levels | Weeks 0 to Week 24 on Step 2
Change in plasma HIV-1 RNA viral load as measured by single copy assay (SCA) | Weeks 0 to Week 24 on Step 2
Change in intact proviral DNA levels (IPDA) | Weeks 0 to Week 24 on Step 2
HIV-1-specific T-cell responses to the conserved regions present in the vaccines as measured by IFN-γ ELISPOT - total frequency and breadth (number of recognized peptide pools out of 10). | Week 0 to Week 24 on Step 2
Change in soluble markers of systemic inflammation and immune activation: sCD163 (pg/mL) | Weeks 0 to Week 24 on Step 2
Change in soluble markers of systemic inflammation and immune activation: sCD14 (pg/mL) | Weeks 0 to Week 24 on Step 2
Change in soluble markers of systemic inflammation and immune activation: IL-6 (pg/mL) | Weeks 0 to Week 24 on Step 2
Change in soluble markers of systemic inflammation and immune activation: sTNFαR (pg/mL) | Weeks 0 to Week 24 on Step 2
Changes in soluble markers of systemic inflammation and immune activation: hsCRP (pg/mL) | Weeks 0 to Week 24 on Step 2
Time to first HIV-1 RNA ≥1000 copies/mL after ATI. | Week 0 to Week 24 on Step 2
Change in HIV-specific CD8+ T-cell-mediated viral inhibition as measured by in vitro virus inhibition assay (VIA) using representative viruses from major HIV-1 clades of group M. | Weeks 0 to Week 24 on Step 2
Occurrence of Medically Attended Adverse Events (MAAEs) | Week 0 on Step 1 to 12 months following the last dose of study vaccination
Occurrence of Adverse Events of Special Interest (AESIs) | Week 0 on Step 1 to 12 months following the last dose of study vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Riddler, MD, MPH, Study Chair — University of Pittsburgh
Locations (12):
- United States (10):
  - University of California, San Diego AntiViral Research Center CRS, San Diego, California
  - Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics CRS, St Louis, Missouri
  - Columbia Physicians & Surgeons CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas
- Brazil (2):
  - Instituto de Pesquisas em AIDS do Rio Grande do Sul - IPARGS CRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.
URL: http://actgnetwork.org/submit-a-proposal/